CLINICAL TRIAL: NCT01659229
Title: Fluoroscopic Analysis Comparing the Dynamic Flexion of 2 Different Knee Arthroplasty Implants
Brief Title: Fluoroscopic Analysis of PFC CR 150 Versus Standard PFC CR Total Knee Arthroplasty Implants in Deep Flexion
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Singapore General Hospital (Other)
Collaborators: DePuy International (Industry)
Responsible Party: Sponsor
Other Study IDs: 63214040
Record Dates: First submitted 2012-08-03; First posted 2012-08-07 (Estimated); Last update posted 2012-08-20 (Estimated); Status verified 2012-08

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PFC CR 150 total knee implant: Study group implant: PFC CR 150 Control group implant: PFC CR standard
- PFC CR Standard: study group implant: PFC CR 150 control group implant: PFC CR Standard

SUMMARY:
The investigators are comparing the range of movements the knees of patients who had total knee replacement surgery for knee osteoarthritis. In the study arm, the implant used was a Sigma Cruciate Retaining (CR) Press Fit Condylar (PFC) 150, which is a high flexion knee system designed to combine function with wear resistance. It can accommodate up to 150 degrees of knee flexion. In the cohort arm, the implant used was the standard Sigma CR which can accommodate up to 120 degrees of flexion.

DETAILED DESCRIPTION:
Both sets of patients will undergo routine post-operative follow up in clinic. The study involves patients who had their surgery more than 2 years ago. We assess their range of movement using fluoroscopy. They are asked to perform lunges, squats and climbing up and down 3 steps. The fluoroscopic images are then analysed to assess their individual range of movements.

ELIGIBILITY:
Inclusion Criteria:

* All patients who underwent total knee replacement surgery who received either the PFC CR 150 knee implants or the PFC CR standard knee implant
* Surgery more than 2 years
* Able to walk, climb stairs

Exclusion Criteria:

* Knee stiffness with less than 100 degrees of knee range of movement
* Patients who required revision surgery
* Patients who received an all polyethylene tibial insert
* Patients who received rotating platform tibial tray

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent total knee replacement surgery who received either the PFC CR 150 knee implants or the PFC CR standard knee implant
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2011-10; Primary Completion 2012-07 (Actual); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Flexion-extension range of movement of operated knee | 2 years after their total knee replacement surgery
  Fluoroscopic studies are done as patient perform lunges, squats and climb up and down stairs.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Seng Jin Yeo, MBBS FRCS, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore, Singapore

REFERENCES:
- [Background] Nicholls RL, Schirm AC, Jeffcote BO, Kuster MS. Tibiofemoral force following total knee arthroplasty: comparison of four prosthesis designs in vitro. J Orthop Res. 2007 Nov;25(11):1506-12. doi: 10.1002/jor.20438. PMID 17568418